CLINICAL TRIAL: NCT05163132
Title: Correlation Between Shear-wave Elastography and CT in Diffuse Liver Disease
Brief Title: Shear-wave Elastography Diffuse Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab Mohamed, Principal Investigator, Assiut University
Other Study IDs: Fibroscan
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Chronic Hepatic; Chronic Liver Disease and Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Shearwave elastography — Shear wave elastography is an ultrasound applied technique used to measure tissue stiffness as a result of a disease. So, it can be used to evaluate liver stiffness as a result of liver cirrhosis

SUMMARY:
The aim of this study is to correlate between quantitative results of shear wave elastography and CT picture in diffuse liver disease, including liver cirrhosis.

DETAILED DESCRIPTION:
Many pathophysiological processes can lead to diffuse parenchymal liver diseases and the end-result of all chronic liver diseases is healing by fibrosis and regeneration. Liver fibrosis is a slowly progressing disease in which healthy liver tissue is replaced with scar tissue ended with liver cirrhosis, with a variety of causes, including viral, drug induced, autoimmune, cholestatic, and metabolic diseases.

Liver biopsy is the gold standard but limited due to its invasiveness, sampling error, and intra- and interobserver variability. Non-invasive tests are preferred in the management of chronic liver diseases. Several serum tests for liver function and markers of liver fibrosis are available and have moderate sensitivity and specificity; however, they are confounded by a wide range of extra-hepatic diseases.

Currently, several methods are available for assessing hepatic fibrosis and progression of fibrogenesis including scintigraphy, magnetic resonance diffusion weighted imaging, and magnetic resonance spectroscopy could differentiate between cirrhosis or severe fibrosis and normal liver. However, an accurate staging of fibrosis or diagnosis of mild fibrosis was often not achievable. Shear-wave elastography (SWE) is a real-time freehand ultrasonography-based elastography method for liver stiffness measurement.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes are included: patients who diagnosed to had chronic liver diseases with or without present hepatic focal lesions.

Exclusion Criteria:

* Lactating and pregnant women
* Patients known to had high serum creatinine

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients who diagnosed to had chronic liver diseases with or without present hepatic focal lesions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Shearwave elastography (SWE) of the liver | 1 week
  Analyze the correlation between SWE of liver and with computed tomography findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdeltawab, MD, Study Director — Assiut; Hayam M Abd El-hakeem, Principal Investigator — Assiut University; Eman Abo El-hamd, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boll DT, Merkle EM. Diffuse liver disease: strategies for hepatic CT and MR imaging. Radiographics. 2009 Oct;29(6):1591-614. doi: 10.1148/rg.296095513. PMID 19959510
- [Result] Lingala S, Ghany MG. Natural History of Hepatitis C. Gastroenterol Clin North Am. 2015 Dec;44(4):717-34. doi: 10.1016/j.gtc.2015.07.003. Epub 2015 Aug 25. PMID 26600216
- [Result] Wilkins T, Akhtar M, Gititu E, Jalluri C, Ramirez J. Diagnosis and Management of Hepatitis C. Am Fam Physician. 2015 Jun 15;91(12):835-42. PMID 26131943
- [Result] Ferraioli G, Tinelli C, Dal Bello B, Zicchetti M, Filice G, Filice C; Liver Fibrosis Study Group. Accuracy of real-time shear wave elastography for assessing liver fibrosis in chronic hepatitis C: a pilot study. Hepatology. 2012 Dec;56(6):2125-33. doi: 10.1002/hep.25936. Epub 2012 Aug 31. PMID 22767302